CLINICAL TRIAL: NCT01593761
Title: Phase 2a, Repeated-dose, Open-label, Single-arm Study of CG400549 for the Treatment of Complicated Acute Bacterial Skin and Skin Structure Infection (cABSSSI) Caused by Methicillin-resistant Staphylococcus Aureus (MRSA)
Brief Title: Phase 2a Study of CG400549 for the Treatment of cABSSSI Caused by Methicillin-resistant Staphylococcus Aureus
Acronym: CG400549
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CG400549-2-01
Record Dates: First submitted 2012-05-06; First posted 2012-05-08 (Estimated); Results first posted 2022-07-06 (Actual); Last update posted 2022-09-10 (Actual); Status verified 2022-08

CONDITIONS: Skin Infection
Keywords: cABSSSI; MRSA
MeSH Terms: conditions — Cellulitis | interventions — CG 400549

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm for CG400549 (Experimental): All the patients will be administered with CG400549.
  Interventions: Drug: CG400549

INTERVENTIONS:
Drug: CG400549 — 960mg QD at fed state approx 1 hour after meal

SUMMARY:
Primary Objective:

To make a preliminary assessment of the efficacy of CG400549 (960 mg daily) in subjects with cABSSSI (major cutaneous abscesses) due to MRSA.

Secondary Objective(s):

* To assess the pharmacokinetics of CG400549 (960 mg daily) in subjects with cABSSSI due to MRSA
* To explore the in vitro susceptibility of cABSSSI-related bacteria to CG400549.
* To assess the safety of multiple doses of CG400459

DETAILED DESCRIPTION:
This will be an open-label, exploratory study to evaluate the safety, pharmacokinetics, and efficacy of CG400549, daily for 10 to 14 days, in subjects with cABSSSI (major cutaneous abscesses) due to MRSA. All subjects will receive active treatment.

Subjects will begin study treatment upon confirmation of clinical eligibility (ie, confirmation of MRSA infection is not required pretreatment). Subjects who begin treatment with CG400549 and are subsequently not found to have S. aureus infection will be discontinued from study treatment, treated as appropriate for the identified pathogen(s), and followed for safety. These subjects will be included in the safety analyses but not in the primary efficacy analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of major cutaneous abscess suspected or confirmed to be caused by a MRSA.
2. Signs and symptoms should include at least 2 of the following: purulent drainage or discharge, erythema, fluctuance, heat or localized warmth, edema/induration, pain or tenderness to palpation

Exclusion Criteria:

1. Prior systemic or topical antibacterial therapy
2. Severe sepsis or refractory shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S. Overcash, MD, Principal Investigator — eStudysite
Locations (1):
- eStudysite, La Mesa, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with complicated acute bacterial skin and skin structure infection were recruited. Study was conducted from June 2012 to October 2012 at 1 site in the United States.
Groups:
- Subjects Received CG400549, MITT: All enrolled subjects who received any amount of study drug and was equivalent to the safety population.
Period: Overall Study
Arm/Group | Subjects Received CG400549, MITT
Started | 20
Completed | 12
Not Completed | 8
Not completed — Lost to Follow-up | 1
Not completed — culture negative for MRSA at baseline | 5
Not completed — positive for hepatitis C virus | 1
Not completed — secondary cellulitis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Subjects Received CG400549, MITT
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.2 (13.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Status of Subject's Clinical Responses
Description: Stable/improving infection, as defined by the Investigator assessment, was defined as cessation of the spread of the redness, edema, and/or induration of the lesion or reduction in the size (length, width, and shortest distance from the peripheral margin of the abscess) of redness, edema, and/or induration and absence of fever (< 37.7 °C)
Time Frame: Early Clinical Evaluation (ECE, 48 to 72 hours after enrollment)
Population: Among 20 participated subjects, 11 subjects had confirmed MRSA and qualified for the mMITT population
Measure: Number; unit: participants
Groups:
- Subjects Proven MRSA, mMITT: The primary population for evaluation of the primary endpoint and comprised all MITT subjects who had confirmed MRSA
Arm/Group | Subjects Proven MRSA, mMITT
Number analyzed (Participants) | 11
participants
  Stable/ Improving Infection | 10
  No Stable/ Improving Infection | 1

2. Secondary Outcome: Status of Subject's Clinical Response
Description: 1. Clinical cure was defined as absence of fever (< 37.7°C); presence of granulation or wound healing; resolution of pain; and decreased or resolved erythema, edema,induration, and color. Ulceration could persist, but lesions had to appear non-infected to be defined as clinical cure.
  2. Clinical improvement was defined as moderate resolution of 2 or more clinical symptoms.
  3. clinical failure was defined as persistence or progression of baseline signs and symptoms of cABSSSI, development of new signs and symptoms consistent with Gram-positive infection, or inability to complete the study because of AEs
Time Frame: End of Treatment (EOT, 10-14 days after beginning treatment) and Test of Cure (TOC, 21-28 days after beginning treatment)
Population: Among 11 mMITT population who had proven MRSA , 2 subjects had major protocol violations, yielding 9 subjects for CE population
Measure: Number; unit: participants
Groups:
- Subjects Proven MRSA, CE: Primary population for assessment of clinical cure and was defined separately for the EOT and TOC visits.
  The mMITT subjects who did not have major protocol violations and received at least 80% of the planned dose of CG400549 were candidates for the CE population.
  1. CE subjects at EOT who met the above criteria and had a clinical lesion assessment at the EOT visit.
  2. CE subjects at TOC who met the above criteria and had a clinical lesion assessment at the TOC visit.
Arm/Group | Subjects Proven MRSA, CE
Number analyzed (Participants) | 9
participants
  Clinical Cure at EOT | 8 [51.8 to 99.7]
  Clinical Improvement at EOT | 1 [66.4 to 100]
  Clinical Failure at EOT | 0
  Clinical Cure at TOC | 9
  Clinical Improvement at TOC | 0
  Clinical Failure at TOC | 0

3. Secondary Outcome: Status of Subject's Microbial Eradication Response
Description: 1. Microbial eradication was defined by culture (complete absence of all infecting organisms identified at baseline) or presumed because of an absence of clinical symptoms.
  2. Microbiological Persistence was defined as the presence of one or more of the original infecting organisms on the TOC culture or as the absence of cultures in case of clinical failure.
  3. Microbiological Recurrence was defined as the presence on the final culture of an original infecting organism whose eradication had been either documented or presumed a the end of therapy.
Time Frame: as for outcome 2
Population: The ME group was not analyzed because the appropriate post-treatment skin culture data were not accessible due to the improvement of infected lesion.
Groups:
- Subjects Proven MRSA, ME: The primary population for assessment of microbial eradiation and was defined separately for the EOT and TOC visits.
  The mMITT subjects who did not have major protocol violations and received at least 80% of the planned dose of CG400549 were candidates for the ME population.
  1. ME subjects at EOT who met the above criteria and had an interpretable culture for microbial response at EOT.
  2. ME subjects at TOC who met the above criteria and had an interpretable culture for microbial response at TOC.
Arm/Group | Subjects Proven MRSA, ME
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Summary of Adverse Events
Description: Treatment-Emergent Adverse Event (TEAE) are those that
  1. Emerging during treatment, having been absent pre-treatment or
  2. Reemerge during treatment, having been present at baseline but stopped prior to treatment or
  3. Worsen in severity during treatment relative to the pre-treatment state, when the adverse event is continuous.
Time Frame: From time of signing the informed consent to Test of Cure (TOC, 21-28 days after after beginning treatment)
Measure: Number; unit: participants
Groups:
- Subjects Received CG400549, MITT: All enrolled subjects who receive any amount of study drug and was equivalent to the safety population.
- Subjects Proven MRSA, mMITT: The mMITT population was the primary population for evaluation of the primary endpoint and comprised all MITT subjects who had confirmed MRSA
Arm/Group | Subjects Received CG400549, MITT | Subjects Proven MRSA, mMITT
Number analyzed (Participants) | 20 | 11
participants
  Treatment-Emergent Adverse Event (TEAE) | 13 | 10
  Severe TEAE | 0 | 0
  Treatment-Related TEAE | 7 | 5
  Severe Treatment-Related TEAE | 0 | 0
  TEAE with outcome of death | 0 | 0
  TEAE leading to withdrawal of study medic | 0 | 0
  Serious Adverse Event | 0 | 0

5. Secondary Outcome: Mean Plasma Concentration-time Profile of CG400549
Description: The concentrations of CG400549 in plasma collected at each point were analyzed and calculated for its mean plasma concentration.
Time Frame: Day 1 predose, Day 1 1hour, Day 1 2hour, Day 1 4hour
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Subjects Proven MRSA, mMITT: MITT subjects who had confirmed MRSA
Arm/Group | Subjects Proven MRSA, mMITT
Number analyzed (Participants) | 20
ng/mL
  Day 1 predose | 32.921 (101.5)
  Day 1 1hour | 426.921 (488.5)
  Day 1 2hour | 1,366.159 (1028.8)
  Day 1 4hour | 1,618.997 (782.3)

ADVERSE EVENTS:
Time Frame: Serious Adverse Event(SAE) was reported from the time of signing the informed consent, and AE is recorded from the time of the first dose of study drug. AEs and SAEs were recorded until subject's last visit (TOC, day 21-28 after enrollment).
Arm/Group | Subjects Proven MRSA, mMITT | Subjects Received CG400549, MITT
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/20
Other Adverse Events (participants affected / at risk) | 10/11 | 13/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Subjects Proven MRSA, mMITT (N=11) | Subjects Received CG400549, MITT (N=20)
infection (Infections and infestations) | 2 | 2
subcutaneous abscess (Infections and infestations) | 1 | 2
amylase increased (Investigations) | 1 | 2
lipase increased (Investigations) | 1 | 3
tachycardia (Cardiac disorders) | 2 | 2
cellulitis (Infections and infestations) | 1 | 1
impetigo (Infections and infestations) | 1 | 1
injection site cellulitis (Infections and infestations) | 1 | 1
pharyngitis streptococcal (Infections and infestations) | 1 | 1
urinary track infection (Infections and infestations) | 1 | 1
upper respiratory tract infection (Infections and infestations) | 1 | 1
diarrhoea (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
vomiting (Gastrointestinal disorders) | 1 | 1
pyrexia (General disorders) | 2 | 2
injection site reaction (General disorders) | 1 | 1
headache (Nervous system disorders) | 2 | 2
ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
muscle strain (Injury, poisoning and procedural complications) | 1 | 1
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 | 1
abnormal dreams (Psychiatric disorders) | 1 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
rash (Skin and subcutaneous tissue disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than or equal to 60 days but less than or equal to 120 days from the time submitted to the sponsor for review.

The sponsor can request to remove any confidential information (other than study results).